CLINICAL TRIAL: NCT00613340
Title: Randomized Study Comparing the Accuracy and Specificity of Cervical Facet Medial Branch Blocks With 0.25 ml and 0.5 ml of Local Anesthetic
Brief Title: The Specificity of Cervical Facet Medial Branch Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Army Regional Anesthesia and Pain Management Initiative (U.S. Federal Agency)
Responsible Party: Walter Reed Dept. of Clinical Investigation, Marty Green
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA-20008-A
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Neck Pain; Cervical Facet Arthropathy
Keywords: Cervical pain; Zygapophysial joint; Specificity
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cervical medial branch blocks with 0.25 ml of injectate
  Interventions: Procedure: Cervical medial branch blocks
- 2 (Experimental): Cervical medial branch blocks with 0.5 ml of local anesthetic and contrast
  Interventions: Procedure: Cervical medial branch blocks

INTERVENTIONS:
Procedure: Cervical medial branch blocks — Cervical medial branch blocks done with 0.25 ml of local anesthetic and contrast
  Arms: 1
Procedure: Cervical medial branch blocks — Cervical medial branch blocks with 0.5 ml of local anesthetic and contrast
  Arms: 2

SUMMARY:
Cervical facet arthropathy is a common cause of chronic neck pain. The "gold standard" for diagnosis is either blocking the facet joints, or more commonly blocking the medial branch nerves that innervate the joints. However, many studies have found a high false-positive rate when the nerves are blocked using 0.5 ml of local anesthetic. We will randomize patients to receive either cervical facet medial branch blocks with 0.25 ml of local anesthetic and contrast, or 0.5 ml. We will then do a CT scan to determine the accuracy and specificity of each block. Our hypothesis is that using the higher volume (0.5 ml) might be responsible for the high false-positive rate.

DETAILED DESCRIPTION:
Inclusion criteria: Dept. of Defense beneficiaries > 18 years of age; neck pain > 3 months duration; cervical paraspinal tenderness Exclusion criteria: Radicular signs or symptoms; use of anticoagulants or bleeding disorder.

Outcome measures: The number of blocks whereby the contrast bathes the target nerve; the number of blocks whereby the contrast spreads to the medial branch nerve at the adjacent spinal level; the number of times the contrast diffuses into the intervertebral foramen or epidural space. We will also compare pain relief over 8 hours following the block between both volumes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Chronic neck pain > 3 months
* Paraspinal tenderness

Exclusion Criteria:

* Absence of radicular symptoms
* No bleeding diathesis
* Contrast allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of injections | Immediately after nerve blocks.

SECONDARY OUTCOMES:
Pain relief after nerve blocks | 8 hours after blocks

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Dreyfuss P, Schwarzer AC, Lau P, Bogduk N. Specificity of lumbar medial branch and L5 dorsal ramus blocks. A computed tomography study. Spine (Phila Pa 1976). 1997 Apr 15;22(8):895-902. doi: 10.1097/00007632-199704150-00013. PMID 9127924
- [Result] Lord SM, Barnsley L, Bogduk N. The utility of comparative local anesthetic blocks versus placebo-controlled blocks for the diagnosis of cervical zygapophysial joint pain. Clin J Pain. 1995 Sep;11(3):208-13. doi: 10.1097/00002508-199509000-00008. PMID 8535040
- [Derived] Cohen SP, Strassels SA, Kurihara C, Forsythe A, Buckenmaier CC 3rd, McLean B, Riedy G, Seltzer S. Randomized study assessing the accuracy of cervical facet joint nerve (medial branch) blocks using different injectate volumes. Anesthesiology. 2010 Jan;112(1):144-52. doi: 10.1097/ALN.0b013e3181c38a82. PMID 19996954